CLINICAL TRIAL: NCT03458013
Title: Exploring Psychosocial Outcomes in Hand Therapy
Brief Title: Psychosocial Outcomes in Hand Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Abbott Medical Devices (Industry); California Foundation for Occupational Therapy (Other)
Responsible Party: Principal Investigator, Shawn Roll, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS-17-00935
Record Dates: First submitted 2018-02-01; First posted 2018-03-08 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hand Injuries
Keywords: Mindfulness; Complementary Medicine; Integrative Health; Hand Therapy
MeSH Terms: conditions — Hand Injuries | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: We are using a 2-cohort, nonrandomized comparative design focused on assessing feasibility and acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation plus Hand Therapy (Experimental): Participants will be recruited from patients suffering from a traumatic injury who are entering hand therapy at a community based clinic in the Los Angeles area.
  Interventions: Behavioral: Mindfulness Meditation
- Standard Care in Hand Therapy (No Intervention): Participants will be recruited from patients suffering from a traumatic injury who are entering hand therapy at a community based clinic in the Los Angeles area.

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Guided using an mp3 player and noise cancelling headphones, participants will be led through a series of mindfulness meditations lasting approximately 20 minutes each.
  Arms: Mindfulness Meditation plus Hand Therapy

SUMMARY:
Rationale: there is a need for psychosocial symptom management in hand therapy which has been understudied. Mindfulness-based interventions are used to address psychosocial symptoms in other settings such as chronic injury but have yet to be implemented or explored for patients in acute outpatient rehabilitation.

Intervention: a supplemental mindfulness-based intervention (MBI) will be provided to the experimental group while the control group will receive standard care. The MBI will begin with an explanation of the purpose of a mindfulness, how mindfulness relates to hand therapy, and lead to a 20-minute guided meditation using an audio recording.

Objectives: to establish the feasibility of providing a MBI in hand therapy and evaluate preliminary effects of the MBI on patients' stress, anxiety, and depression.

Population: adult patients at an outpatient hand therapy clinic in the Los Angeles area who have received a traumatic injury (e.g., tendon laceration, compound fracture, finger amputation).

Methodology: the study will use a mixed-methods, non-randomized, 2-group, comparative trial design with 40 participants in total. Quantitative data on psychosocial outcomes, including salivary cortisol, will be collected once a week for 4 weeks while patients are attending hand therapy and qualitative interviews will be conducted at the end of the study.

Study arms: the experimental group (n = 20) will receive the MBI just before regularly scheduled standard care visits. The control group (n = 20) will receive only standard care.

Outcomes: this pilot study will be used to inform a future fully powered trial on mindfulness-based interventions in hand therapy. Feasibility and preliminary psychosocial effects of MBIs will be evaluated and used to inform future work.

Analysis: (1) A repeated measures ANOVA for intervention group, time, and time by intervention group effects on the psychosocial outcomes (i.e., Cortisol, Anxiety, Depression, and Pain Catastrophizing). (2) A descriptive qualitative process will be used to analyze themes in participant interview responses.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old; newly entering hand therapy, having a diagnosis of distal radius fracture, flexor tendon injury and repair, extensor tendon injury and repair, tramatic finger amputation, or other traumatic injury; established therapy plan of care lasting at least 4 weeks; able to read and with in English; with regular access to a computer.

Exclusion Criteria:

* diagnosed with a severe mental illness; currently an expert in mindfulness practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Salivary Cortisol Across 4 weeks | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Cortisol is a bio-marker for stress (Aardal & Holm, 1995). Normal values in healthy adults are sensitive to time of day, but range from 3.5 to 27.0 nmol/l in the morning. Higher salivary cortisol levels are an indicator of higher levels of stress.

SECONDARY OUTCOMES:
Change in Baseline State Anxiety Across 4 weeks | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  The State-Trait Anxiety Inventory: State subscale (Spielberger, Vagg, Barker, Donham, & Westberry, 1980) is scored positively (higher scores equate to higher anxiety) with a minimum score of 20 and a maximum score of 80. Normative data for this scale indicates that a cut point score of 40 and above is considered clinically relevant.
Change in Baseline Depression Across 4 weeks | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Center for Epidemiologic Studies - Depression scale (CES-D; Radloff, 1977), is a 20-item depression scale that is positively scored (higher scores equate to higher depression) ranging from 0 to 60. It is intended for use with the general population with a conservative off is score being greater than 16.
Change in Baseline Pain Catastrophizing Baseline Across 4 weeks | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995) measures an individual's exaggerated negative psychological response to pain or the anticipation of pain. The scale is scored positively across 13 total items composing 3 subscales: rumination, magnification, and helplessness. These subscales are added together to get the total score from 0 to 52. The middle 50% of scores on this scale fall between 10 and 30 points.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Roll, PhD, Study Chair — University of Southern California; Mark E Hardison, MS, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - St. Jude Centers for Rehabilitation & Wellness, Brea, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aardal E, Holm AC. Cortisol in saliva--reference ranges and relation to cortisol in serum. Eur J Clin Chem Clin Biochem. 1995 Dec;33(12):927-32. doi: 10.1515/cclm.1995.33.12.927. PMID 8845424
- [Background] Spielberger CD, Vagg PR, Barker LR, Donham GW, Westberry LG. The factor structure of the State-Trait Anxiety Inventory. In CD Spielberger & IG Sarason (Eds.), Stress and anxiety (pp. 244-279). Washington, DC: Hemisphere; 1980.
- [Background] Radloff, LS. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement 1(3): 385-401, 1977.
- [Background] Sullivan MJ, Bishop SR, Pivik J. The pain catastrophizing scale: Development and validation. Psychological Assessment 7(4): 524 - 532, 1995.